CLINICAL TRIAL: NCT01320605
Title: TRIAL OF COMPASSIONATE USE OF HP802-247 TO TREAT VENOUS LEG ULCERS IN SUBJECTS WHO HAVE FAILED MULTIPLE OTHER HEALING TECHNOLOGIES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: David Eisenbud, MD, Overlook Hospital Wound Healing Program
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E001
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly HP802247 treatment (Experimental)
  Interventions: Biological: Weekly wound spray with components 1 and 2 of the compound HP802-247

INTERVENTIONS:
Biological: Weekly wound spray with components 1 and 2 of the compound HP802-247 — Weekly spray with HP802-247

SUMMARY:
Compound HP802-247 comprises two topical sprays, administered sequentially right after another; these deliver a suspension of fibroblasts and keratinocytes to the wound surface. HP802-247 is the subject of a larger Phase 2 multi-center trial for treating venous leg ulcers. The present study will enroll up to five patients who are suffering venous leg ulcers, have failed a prolonged course of standard wound therapy and one or more advanced technologies, but who would not qualify for the Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (duration greater than six months) open wound that has been diagnosed as a venous leg ulcer on the basis of consultation with a vascular surgeon and/or venous ultrasound evaluation
* Patient has been under continuous care at the Overlook Hospital Wound Healing Program for at least four months for treatment of the study lesion(s)
* Total study wound surface area greater than or equal to 12 cm2, but less than 48 cm2
* Wounds must have failed to heal despite the patient's compliance with elevation, compression and regular debridement, as well as at least one advanced wound therapy (for example, bioengineered dressing such as Oasis® or MatriStem®, low-frequency ultrasound, or cultured skin substitute (Apligraf®, Dermagraft®)
* Patient has no reasonable likelihood of healing with additional attempts to treat with FDA-approved products and treatments

Exclusion Criteria:

* Patients eligible to participate in a Healthpoint sponsored clinical study of HP802-247 trial (IND 13,900)
* Patients who have been previously treated with HP802-247
* Women of child-bearing potential
* Patients who are allergic to any of the components of HP802-247

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete wound closure during the treatment period | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Overlook Hospital Wound Healing Program, Summit, New Jersey, United States